CLINICAL TRIAL: NCT06701604
Title: Comparative Differences of Amino Acid Appearance with Milk Protein Ingestion with and Without Probiotic Supplementation
Brief Title: Changes in Amino Acid Absorption After Adding a Probiotic to an Acute Protein Feeding
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Archer-Daniels-Midland Company (Industry)
Collaborators: University of Mary Hardin-Baylor (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: PCTB202104D
Record Dates: First submitted 2024-11-20; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Amino Acid Absorption; Probiotic
MeSH Terms: interventions — Milk Proteins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Milk Protein + Probiotic (Experimental): Arm receiving investigational product (probiotic) in the form of a capsule with a dose of 1B Colony Forming Unit (CFU) per day + a 25-gram dose of milk protein concentrate given daily for 3 weeks
  Interventions: Dietary Supplement: Single Strain Probiotic + Milk Protein
- Milk Protein + Placebo (Placebo Comparator): Arm receiving placebo matching investigational product + a 25-gram dose of milk protein concentrate given daily for 3 weeks
  Interventions: Dietary Supplement: Placebo + Milk Protein

INTERVENTIONS:
Dietary Supplement: Single Strain Probiotic + Milk Protein — • Both conditions matched flavor, color, and serving size
  Arms: Milk Protein + Probiotic
Dietary Supplement: Placebo + Milk Protein — • Both conditions matched flavor, color, and serving size
  Arms: Milk Protein + Placebo

SUMMARY:
The purpose of this study is to examine the rate and concentration of amino acid absorption after a three-week pattern of milk protein supplementation with and without the addition of a single strain probiotic.

DETAILED DESCRIPTION:
The study will be conducted using a randomized, double-blind, crossover study design. Thirty healthy men and women between 18 - 35 years of age will be recruited to participate in this study. Two supplementation protocols that each span three weeks will be completed and separated with a washout period of three weeks. Participants will be assigned in a randomized, double-blind, crossover fashion to ingest a single daily 25-gram dose of a powder milk protein and placebo or a single daily 25-gram dose of a powder milk protein plus a single strain probiotic. Upon arrival for each study visit, participants will have their resting heart rate, blood pressure, body mass, height, and body composition measured. On the day of experimental testing, subjects will arrive to the laboratory in a fasted state. Subjects will rest semi-supine for multiple blood sampling. Following baseline sampling, participants will ingest their respective supplement plus a standard bolus of milk protein (powder form, mixed with 12 fl oz of cold water). Thereafter, blood samples will be taken at 30, 60, 90, 120, 180, and 240 minutes post-ingestion. Study participants will be provided an additional three-week supply of the alternative treatment to begin after observing a three-week washout. After three weeks of supplementation, study participants will return to the laboratory for their remaining testing visit.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be male or female between the ages of 18-35 years;
* Participants have not been consuming any nutritional supplements for the preceding 6-week period;
* Participants have not been consuming any ergogenic aids for the preceding 6-week period;
* Participant has provided written and dated informed consent to participate in the study;
* Participant is willing and able to comply with the protocol;
* Participant is apparently healthy and free from disease, as determined by a health history questionnaire;

Exclusion Criteria:

* Participant is allergic to any ingredient in the nutritional supplement or placebo;
* Participant is not pregnant or trying to become pregnant, nor breast feeding;
* Participant reports any unusual adverse events associated with this study that in consultation with the study investigators or their doctor recommends removal from the study;
* Participant currently ingests nicotine or has quit within the last 6 months;

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12-02 (Estimated); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Rate of amino acid absorption | Day 0, Day 22, Day 65
  To determine if the addition of a probiotic to milk protein ingestion changes the rate (in minutes) to which amino acids are absorbed into our bloodstream.
Concentration of amino acid absorption | Day 0, Day 22, Day 65
  To determine if the addition of a probiotic to milk protein ingestion changes the extent (concentration in millimoles/Liter) to which amino acids are absorbed into our bloodstream.

SECONDARY OUTCOMES:
Comprehensive metabolic panel | Day 0, Day 22, Day 65
  Comprehensive metabolic panel will be assessed pre vs. post supplementation across the two treatment groups for blood safety data.
  • All measures are assessed by blood or serum assay analysis
Blood CBC panel | Day 0, Day 22, Day 65
  Blood CBC panel will be assessed pre vs. post supplementation across the two treatment groups for blood safety data.
  • All measures are assessed by blood or serum assay analysis

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Mary Hardin-Baylor, Belton, Texas, United States

IPD SHARING:
Plan to Share IPD: No